CLINICAL TRIAL: NCT01971125
Title: Left Ventricular DYsfunction in DiAbetes
Acronym: DYDA
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: G 107
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2013-10

CONDITIONS: Diabetes Mellitus, Type 2; Heart Diseases; Left Ventricular Dysfunction
Keywords: Diabetes Mellitus, Type 2; Heart Diseases; Left Ventricular Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Patients with:
  * diabetes mellitus type 2
  * absence of heart disease previously reported
  * age >45 years
  * Informed Consent
  Patients without:
  * presence of heart disease previously reported
  * diabetes type 1
  * serious systemic disease, with an expected lifetime lower than 2 years
  * no willingness to participate to the screening
  * inadequate compliance to study procedure
  * participation to other study

SUMMARY:
The purpose of this study is to evaluate the prevalence, during the enrolment, of Left Ventricular Dysfunction diastolic and/or systolic in patients with diabetes mellitus type 2 without known or documented heart disease history and recognize its predictive clinical, biohumoral and with non-invasive techniques parameters.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 2
* absence of heart disease previously reported
* age >45 years
* Informed Consent

Exclusion Criteria:

* presence of heart disease previously reported
* diabetes type 1
* serious systemic disease, with an expected lifetime lower than 2 years
* no willingness to participate to the screening
* inadequate compliance to study procedure
* participation to other study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus type 2 without known or documented heart disease history and recognize its predictive clinical, biohumoral and with non-invasive techniques parameters.
Sampling Method: Non-Probability Sample
Enrollment: 970 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of Left Ventricular Dysfunction in patients with type II diabetes | left ventricula dysfunction at enrollment
  To evaluate the prevalence of left ventricular dysfunction (LVD), diastolic or systolic in patients with type II diabetes mellitus in the absence of clinical signs/symptoms of cardiac abnormalities To identify the predictors of LVD

CONTACTS AND LOCATIONS:
Overall Officials: Marco Comaschi, M.D., Study Chair; Andrea di Lenarda, M.D., Study Chair
Locations (14):
- Italy (14):
  - Casa di Cura Pineta del Carso, Duino-Aurisina, Friuli Venezia Giulia
  - A.O.- Univ. Ospedali Riuniti, Trieste, Friuli Venezia Giulia
  - Azienda Servizi Sanitari N°1 Triestina, Trieste, Friuli Venezia Giulia
  - Presidio Ospedaliero, Sanremo, Liguria
  - Ospedali Riuniti, Bergamo, Lombardy
  - Spedali Civili, Brescia, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Ospedale San Paolo, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - IRCCS Policlinico Multimedica, Sesto San Giovanni, Lombardy
  - Ospedale Maggiore, Chieri, Piedmont
  - A.O. Santa Croce e Carle, Cuneo, Piedmont
  - Ospedale Mauriziano, Turin, Piedmont
  - Ospedale Civile, Mirano, Veneto

REFERENCES:
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Cioffi G, Giorda CB, Chinali M, Di Lenarda A, Faggiano P, Lucci D, Maggioni AP, Masson S, Mureddu GF, Tarantini L, Velussi M, Comaschi M; DYDA Investigators. Analysis of midwall shortening reveals high prevalence of left ventricular myocardial dysfunction in patients with diabetes mellitus: the DYDA study. Eur J Prev Cardiol. 2012 Oct;19(5):935-43. doi: 10.1177/1741826711417759. Epub 2011 Jul 28. PMID 21798988
- [Background] Cioffi G, Faggiano P, Lucci D, Di Lenarda A, Mureddu GF, Tarantini L, Verdecchia P, Comaschi M, Giorda CB, Velussi M, Chinali M, Latini R, Masson S, De Simone G; DYDA Investigators. Inappropriately high left ventricular mass in patients with type 2 diabetes mellitus and no overt cardiac disease. The DYDA study. J Hypertens. 2011 Oct;29(10):1994-2003. doi: 10.1097/HJH.0b013e32834acc6d. PMID 21881524
- [Background] Cioffi G, Faggiano P, Lucci D, Maggioni AP, Manicardi V, Travaglini A, Girfoglio D, Masson S, Giorda CB, Velussi M, Di Lenarda A, Verdecchia P, Comaschi M. Left ventricular dysfunction and outcome at two-year follow-up in patients with type 2 diabetes: The DYDA study. Diabetes Res Clin Pract. 2013 Aug;101(2):236-42. doi: 10.1016/j.diabres.2013.05.010. Epub 2013 Jun 24. PMID 23806478
- [Background] Masson S, Latini R, Cioffi G, Urso R, Vago T, Lucci D, Mureddu GF, Tarantini L, Faggiano P, Girfoglio D, Velussi M, Maggioni AP, Giorda CB, Comaschi M; DYDA Investigators. Cardiovascular biomarkers, cardiac dysfunction, and outcomes in patients with type 2 diabetes: a prospective, multicenter study. Diabetes Care. 2013 Sep;36(9):e137-8. doi: 10.2337/dc13-0836. No abstract available. PMID 23970719
- [Result] Giorda CB, Cioffi G, de Simone G, Di Lenarda A, Faggiano P, Latini R, Lucci D, Maggioni AP, Tarantini L, Velussi M, Verdecchia P, Comaschi M; DYDA Investigators. Predictors of early-stage left ventricular dysfunction in type 2 diabetes: results of DYDA study. Eur J Cardiovasc Prev Rehabil. 2011 Jun;18(3):415-23. doi: 10.1177/1741826710389402. Epub 2011 Feb 22. PMID 21450640
- See also: Related Info — http://www.anmco.it/Dyda